CLINICAL TRIAL: NCT06678932
Title: Comparison of Arm Exercise Capacity, Muscle Strength and Daily Living Activities of Patients with Fibromyalgia Syndrome and Healthy Controls
Brief Title: Arm Exercise Capacity, Muscle Strength and Activities of Daily Living in Patients with Fibromyalgia Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-13/115
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fibromyalgia syndrome
- Healthy controls

SUMMARY:
The aim of this study is to compare the upper extremity exercise capacity, muscle strength and activities of daily living of patients with fibromyalgia syndrome and healthy individuals.

ELIGIBILITY:
Inclusion Criteria-fibromyalgia syndrome:

* Being diagnosed with fibromyalgia syndrome
* Being aged 18-65
* Stable use of medication for at least 3 months or longer
* Volunteering to participate in the study

Exclusion Criteria-fibromyalgia syndrome:

* Having comorbidities that may affect physical functions
* Failure to cooperate with tests to be performed
* Presence of exercise test contraindication

Inclusion Criteria-healthy control:

* Being aged 18-65
* Volunteering to participate in the study

Exclusion Criteria-healthy control:

* Having a chronic or systemic disease
* Failure to cooperate with tests to be performed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with fibromyalgia syndrome and healthy individuals will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Upper extremity exercise capacity | 1st day
  This will be evaluated with arm ergometer test.
Muscle strength | 1st day
  Hand grip strength will be measured using a hand grip dynamometer.
Muscle endurance | 1st day
  30 second push-up test will be used, and total number will be recorded.
Activities of daily living | 1st day
  It will be evaluated with the Glittre Activities of Daily Living test, and total time will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Kavalci Kol, Study Chair — Kirsehir Ahi Evran University; Figen Tuncay, Study Chair — Kirsehir Ahi Evran University
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)